CLINICAL TRIAL: NCT01281748
Title: Evaluation Of The Efficacy Of Corticosteroids In Patients With An Acute Exacerbation Of Chronic Obstructive Pulmonary Disease Receiving Ventilator Support
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low rate of enrollment
Sponsor: Hospital Universitario Getafe (Other)
Collaborators: GRANT IP041233 FROM FONDO DE INVESTIGACION SANITARIA (Unknown)
Responsible Party: Inmaculada Alía, Miguel Angel de la Cal and Andrés Esteban, Hospital Universitario de Getafe
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CORTICOSTEROIDS AND ACUTE COPD
Record Dates: First submitted 2011-01-20; First posted 2011-01-24 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2005-05

CONDITIONS: COPD
Keywords: acute exacerbation of COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- methylprednisolone (Experimental)
  Interventions: Drug: intravenous methylprednisolone
- normal saline solution (Placebo Comparator)
  Interventions: Other: intravenous normal saline solution

INTERVENTIONS:
Drug: intravenous methylprednisolone — methylprednisolone 0,5 mg/kg every 6 hours for 72 hours, 0,5 mg/kg every 12 hours on days 4 through 6, 0,5 mg/kg daily for day 7 through day 10
  Arms: methylprednisolone
Other: intravenous normal saline solution — 50 ml of intravenous normal saline solution every 6 hours for 72 hours, 50 ml every 12 hours on days through 6, 50 ml daily for day 7 through day 10.
  Arms: normal saline solution

SUMMARY:
Clinical practice guidelines for the management of chronic obstructive pulmonary disease (COPD) recommend treatment with systemic corticosteroids during acute exacerbations. The results of a Cochrane systematic review show that treatment with systemic corticosteroids improves lung function over the first 72 hours of an exacerbation of COPD but the effect on other outcomes, particularly length of hospital stay, is unclear, so further research should be directed at determining the risk-benefit ratio, particularly those at high risk of developing adverse drug reactions. In critically ill patients, corticosteroid treatment is a risk factor of infections, hyperglucemia and critical-illness neuromuscular abnormalities, and these conditions are associated with an increased morbidity and mortality. The effect of treatment with systemic corticosteroids in COPD patients with acute exacerbation requiring mechanical ventilation has not been evaluated investigated so it is unknown if the corticosteroids could reduce the duration of mechanical ventilation and the length of intensive care unit (ICU) stay or if, on the contrary, the development of adverse events could lead to a longer time on mechanical ventilation and ICU stay.

PRIMARY OBJECTIVES: To evaluate the effect of corticosteroids on the duration of mechanical ventilation, the length of ICU stay, the need for tracheal intubation in patients treated with non-invasive mechanical ventilation. To evaluate the frequency of adverse events: secondary infections, pneumonia, arterial hypertension, hyperglucemia, gastrointestinal bleeding, and critical-illness neuromuscular abnormalities. DESING: Multicenter, prospective, randomized, double blind, placebo-controlled clinical trial.The treatment group will receive intravenous methylprednisolone for 10 days and the control group will receive isotonic saline solution.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18 years) admitted to participating ICUs with:

  1. Primary diagnosis of COPD exacerbation defined as the presence of two or more of the following clinical features: worsening dyspnea, increase in sputum purulence, increase in sputum volume
  2. respiratory failure [pH < 7,35 with a PaCO2 > 45 mm Hg and respiratory rate more than 23 breaths per minute] requiring mechanical ventilation, invasive or non-invasive mechanical ventilation.

Exclusion Criteria:

1. Primary diagnosis of asthma exacerbation.
2. History of asthma or atopy.
3. Use of systemic corticosteroids within the preceding month.
4. Use of systemic corticosteroids for the treatment of COPD exacerbation at the time of ICU admission for more than 24 hours.
5. Clinical or radiological evidence of pneumonia.
6. Uncontrolled left-ventricular failure (patients with evidence of severe heart failure requiring inotropes or vasoactive drugs).
7. Uncontrolled hypertension arterial (systolic pressure > 180 mm Hg or diastolic pressure > 90 mm Hg despite antihypertensive therapy).
8. Uncontrolled diabetes mellitus.
9. Presence of a neuromuscular disease.
10. History of allergy and or adverse reaction to corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2005-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Duration of mechanical ventilation | Participants are followed until ICU discharge
  Time elapsed between tracheal intubation and extubation (in the group of patients treated with invasive mechanical ventilation),or time elapsed between initiation of non-invasive mechanical ventilation and withdrawal of non-invasive mechanical ventilation (in the group of patients successfully treated with non-invasive mechanical ventilation, or time elapsed between initiation of non-invasive ventilation and extubation (in the case of those patients who failed non-invasiev ventilation and required tracheal intubation).
Need for intubation in patients treated with non-invasive mechanical ventilation | Participants are followed until ICU discharge
  Number of patients intubated in the following 48 hours after the initiation of non-invasive mechanical ventilation
Length of ICU stay | Participants are followed until ICU discharge
  Time elapsed between ICU admission and ICU discharge (dead or alive)

SECONDARY OUTCOMES:
ICU mortality | Participants are followed until ICU discharge
  Number of participants who die in the ICU
Length of hospital stay | Participants are followed until hospital discharge
  Time elapsed between hospital admission and hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Getafe, Getafe, Madrid, Spain

REFERENCES:
- [Derived] Alia I, de la Cal MA, Esteban A, Abella A, Ferrer R, Molina FJ, Torres A, Gordo F, Elizalde JJ, de Pablo R, Huete A, Anzueto A. Efficacy of corticosteroid therapy in patients with an acute exacerbation of chronic obstructive pulmonary disease receiving ventilatory support. Arch Intern Med. 2011 Nov 28;171(21):1939-46. doi: 10.1001/archinternmed.2011.530. PMID 22123804